CLINICAL TRIAL: NCT00140959
Title: Antihypertensive Effects of a Fixed-dose Combination of Losartan and Hydrochlorothiazide Plus Amlodipine Versus a Hydrochlorothiazide and Atenolol Combination Plus Amlodipine in Subjects With Ambulatory Systolic Hypertension.
Brief Title: Losartan and HCTZ and Amlodipine vs Atenolol and Amlodipine (0954A-309)(COMPLETED)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0954A-309; 2005_061
Record Dates: First submitted 2005-08-31; First posted 2005-09-01 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Losartan; Duration of Therapy; Hydrochlorothiazide; Amlodipine; Atenolol

INTERVENTIONS:
Drug: MK0954, losartan potassium/Duration of Treatment: 18 weeks
Drug: Comparator: losartan, HCTZ, amlodipine, atenolol/Duration of Treatment: 18 weeks

SUMMARY:
A study to evaluate the effects of combination losartan versus combination atenolol in patients with ambulatory systolic hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Males or females at least 18 years of age who have ambulatory systolic hypertension.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2003-02-01 (Actual); Primary Completion 2004-06-30 (Actual); Study Completion 2004-06-30 (Actual)

PRIMARY OUTCOMES:
Mean daytime ambulatory systolic blood pressure

SECONDARY OUTCOMES:
Ambulatory BP
Pulse pressure
Trough sitting BP
Percentage of patients who reach goal ambulatory systolic BP

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Lacourciere Y, Poirier L, Lefebvre J. Expedited blood pressure control with initial angiotensin II antagonist/diuretic therapy compared with stepped-care therapy in patients with ambulatory systolic hypertension. Can J Cardiol. 2007 Apr;23(5):377-82. doi: 10.1016/s0828-282x(07)70771-7. PMID 17440643